CLINICAL TRIAL: NCT05987592
Title: BE WELL With Migraine: Brain Education and WELLness With Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00079570; R01AT011502 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Migraine
Keywords: Migraine; Migraine without aura; Migraine with aura; behavioral; mind-body; integrative; virtual; online
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura; Behavior | interventions — Health

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment in which one group receives treatment A and the other group receives treatment B
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study PI, statistician, co-investigators, and all personnel who are involved in endpoint assessments, will be blinded.
  In addition, blinded reports will be provided to the Wake Forest Data and Safety Monitoring Board (DSMB) for safety monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Education and WELLness with Migraine Group A (Experimental): 8 weekly virtual sessions plus online platform
  Interventions: Behavioral: Brain Education and WELLness with Migraine Group A
- Brain Education and WELLness with Migraine Group B (Experimental): 8 weekly virtual sessions plus online platform
  Interventions: Behavioral: Brain Education and WELLness with Migraine Group B

INTERVENTIONS:
Behavioral: Brain Education and WELLness with Migraine Group A — Behavioral intervention that involves 8 weekly group virtual sessions with an instructor that may help improve migraine, plus access to an online platform with additional content and learning
  Other Names: Migraine Group A
  Arms: Brain Education and WELLness with Migraine Group A
Behavioral: Brain Education and WELLness with Migraine Group B — Behavioral intervention that involves 8 weekly group virtual sessions with an instructor that may help improve migraine, plus access to an online platform with additional content and learning
  Other Names: Migraine Group B
  Arms: Brain Education and WELLness with Migraine Group B

SUMMARY:
The goal of this randomized clinical trial is to evaluate two different non-drug, virtual treatment options designed to improve the lives of patients with migraine. Both interventions involve 8 weekly sessions and an online platform with additional content and learning. Participants can stay on all their medications during this study. Information from this study may help determine how to better treat migraine.

DETAILED DESCRIPTION:
This study involves 8 weekly virtual sessions & an online platform designed to improve the lives of patients with migraine. Participants from across the United States with migraine may be eligible to participate. This study does not require any in-person visits. All assessments and surveys will be completed virtually and/or online. Participants will independently complete an initial online screen. Participants will attend a scheduled phone or videoconferencing call with a study team member to complete the baseline assessment and learn how to use the online platform. Participants will keep an online daily headache log and complete several online surveys throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with or without aura by with headache frequency of 4-20 days/month
* At least 1 year of migraine
* At least 18 years old
* Able to participate in 8 weekly online classes
* Willingness to complete baseline headache logs
* Headache-related disability (Headache Impact Test (HIT)-6) score >50
* Fluent in English
* Completion of technology onboarding with the online platform
* Pregnant women who are less than or equal to 16 weeks gestation at enrollment are allowed to participate

Exclusion Criteria:

* Major unstable medical/psychiatric condition that could be unsafe for participants or for the group environment.
* Medication overuse headache, with migraine treatment
* Pregnant women who are more than 16 weeks gestation at enrollment
* Unstable migraine treatment at enrollment: any preventive treatment (oral or injectable medication or neuromodulatory device) started within 12 weeks OR acute treatment within 4 weeks to ensure stability
* Unwillingness to maintain stable current medication dosages for study duration
* Failure to complete baseline headache logs
* Heavy alcohol and illicit drug use
* Participation in another intervention clinical trial or one that would interfere in this study
* Experience with stress reduction training (daily meditation practice, regular use of a mindfulness app, or prior experience with MBSR)
* Any, and all other diagnoses or conditions which, in the opinion of the site investigator, would prevent the patient from being a suitable candidate for the study or interfere with the medical care needs of the study participant: COVID-positive test within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Disability assessed using monthly Migraine Disability Assessment (mMIDAS) - Change in Migraine Disability from baseline to 8 weeks | Immediately post-intervention at 8 weeks
  Most frequently used headache disability measure developed by Dr. Richard Lipton that captures both presenteeism and absenteeism. Although originally developed to report the prior 3 months, the monthly MIDAS ("mMIDAS") reduces recall bias and improves validity.

SECONDARY OUTCOMES:
Depression assessed using Patient Health Questionnaire (PHQ-8) Questionnaire - Change in Depression from baseline to 8 weeks | Immediately post-intervention at 8 weeks
  PHQ-8 has equivalent diagnostic depression accuracy as PHQ-9 and will be used to assess depression. PHQ-8 scores range from 0 to 24. Each of the 9 items can be scored from 0 ("not at all") to 3 ("nearly every day"). Cut-points of 5, 10, 15, and 20 represent the thresholds for mild, moderate, moderately severe, and severe depression, respectively.
Pain Catastrophizing quantified using Pain Catastrophizing Scale (PCS) - Change in Pain catastrophizing from baseline to 8 weeks | Immediately post-intervention at 8 weeks
  This 13-item scale quantifies an individual's pain experience. Unlike other scales, this does not require for the person to be in pain while completing it. Patients are asked to rate the degree to which they have any of the thoughts described in the questionnaire using a 5-point Likert scale ranging from 0 (never) to 4 (always). The total score is the sum of the scores for the individual items, and ranges from 0 to 52.
Self-Efficacy assessed with the Headache Management Self-Efficacy Scale (HMSE) - Change in Self-efficacy from baseline to 8 weeks | Immediately post-intervention at 8 weeks
  A 25-item scale that assesses patient's beliefs in their ability to prevent and/or appropriately manage their headaches and headache-related disability; it has been shown to be valid and reliable. This scale consists of 25 items rated on a 7-point scale that ranges from 1 strongly disagree to 7 strongly agree. Total scores range from 0-175, higher scores reflect more self-efficacy.
Disability assessed using monthly Migraine Disability Assessment (mMIDAS) at 20 weeks - Change in migraine disability from baseline to 20 weeks | Post-intervention at 20 weeks
  Most frequently used headache disability measure developed by Dr. Richard Lipton that captures both presenteeism and absenteeism. Although originally developed to report the prior 3 months, the monthly MIDAS ("mMIDAS") reduces recall bias and improves validity.
Disability assessed using monthly Migraine Disability Assessment (mMIDAS) at 32 weeks - Change in migraine disability from baseline to 32 weeks | Post-intervention at 32 weeks
  Most frequently used headache disability measure developed by Dr. Richard Lipton that captures both presenteeism and absenteeism. Although originally developed to report the prior 3 months, the monthly MIDAS ("mMIDAS") reduces recall bias and improves validity.
Anxiety assessed using Generalized Anxiety Disorder-7 (GAD-7) at 8 weeks - Change in anxiety from baseline to 8 weeks | Immediately post-intervention at 8 weeks
  This is a 7-item scale that quantifies and assess the severity of generalized anxiety disorder, over the past 2 weeks - GAD-7 score of 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe)
Quality of Life assessed using Migraine Specific Quality of Life version 2.1 (MSQL v2.1) at 8 weeks | Immediately post-intervention at 8 weeks
  This is a 14-item questionnaire that measures how migraines affect a patient's daily life and is a highly reliable and valid instrument. The raw scores are transformed to a 0-100 scale and higher scores reflect greater quality of life
Migraine frequency using the daily and 7-day recall headache log at 8 weeks - Change in migraine frequency from baseline to 8 weeks | Immediately post-intervention at 8 weeks
  Participants will complete a daily headache log (<10 items) that captures frequency, along with a 7-day recall headache log (<10 items).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Wells, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Cambridge Health Alliance - Center for Mindfulness and Compassion, Cambridge, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to our outcome measures will be included in the IPD Sharing Statement (IPD) sharing plan, in addition to our study protocol, informed consent, and analytic plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and within 12 months of completion of the analysis of study primary aims and ending within 36 months, anonymous and de-identified data will be made available on clinicaltrials.gov so that other investigators can verify or follow-up on the reported analyses.
Access Criteria: Investigators whose proposed use of the data has been approved by an IRB identified for this purpose - For individual participant data meta-analysis - Data will be made available on clinicaltrials.gov